CLINICAL TRIAL: NCT01309672
Title: Abiraterone Acetate Treatment for Prostate Cancer Patients With a PSA of More Than Four Following Initial Androgen Deprivation Therapy Phase II
Brief Title: S1014 Abiraterone Acetate in Treating Patients With Prostate Cancer Who Have Undergone Initial Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000696565; S1014 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; hormone-resistant prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abiraterone acetate + prednisone (Experimental): Abiraterone, 1,000 mg, oral (on an empty stomach at least 2 hours after or 1 hour before eating); to be taken daily
  Prednisone, 5 mg, oral, 5 mg twice daily
  Interventions: Drug: abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: abiraterone acetate — 1,000 mg, oral (on an empty stomach at least 2 hours after or 1 hour before eating); taken daily
Drug: Prednisone — 5 mg, oral, 5 mg twice daily

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Antiandrogen drugs, such as abiraterone acetate, may lessen the amount of androgens made by the body. It may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying the side effects and how well abiraterone acetate works in treating patients with prostate cancer who have undergone initial hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the rate of achieving a prostate-specific antigen (PSA) of ≤ 0.2 ng/mL with abiraterone acetate therapy in men with metastatic prostate cancer with a sub-optimal response to androgen-deprivation therapy (ADT).

Secondary

* To assess the overall survival and objective progression-free survival of this group of patients.
* To assess PSA partial response.
* To evaluate the qualitative and quantitative toxicity of abiraterone acetate.

OUTLINE: This is a multicenter study.

Patients receive abiraterone acetate orally daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients receive androgen blockade with GNRH agonist (goserelin acetate or leuprolide acetate) or a GNRH antagonist (degarelix) per the treating physician and this will be given continuously until evidence of disease progression. Bilateral surgical orchiectomy is also acceptable.

After completion of study therapy, patients are followed up every 3 months for 1 year and then every 6 months for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven diagnosis of adenocarcinoma of the prostate

  * Metastatic (M1) disease as evidenced by soft tissue and/or bony metastases at the time of initiation of androgen-deprivation therapy (ADT)
  * Must have at least one of the following:

    * Visceral disease (liver, lung, other viscera)
    * Bone metastases to sites in either the axial (spine, pelvis, ribs, or skull) and/or the appendicular (clavicle, humerus, or femur) skeleton
    * Distant lymph node disease (e.g., above the aortic bifurcation, etc.)
  * No small cell or neuroendocrine prostate cancer
* Patients must be receiving ADT (e.g., gonadotropin-releasing hormone [GNRH] antagonist, with or without antiandrogen) prior to entering this study

  * Degarelix, a FDA-approved GNRH antagonist, is an acceptable form of ADT
  * Bilateral surgical orchiectomy is also acceptable
* Suboptimal response to ADT induction as defined by the following criteria:

  * Declining PSA (current PSA is less than the PSA prior to starting ADT) that fails to reach 4 ng/mL or below despite continuous ADT

    * PSA of > 4 ng/mL must be observed between 6-12 months after the initiation of ADT
    * Documentation of failure to achieve this PSA of ≤ 4 ng/mL must be within 28 days of registration

      * The PSA must be obtained after any applicable antiandrogen washout period
    * If the PSA is declining or stable (defined as a PSA rise ≤ 0.1 ng/mL from nadir) and the patient is on an antiandrogen, they must remain on the antiandrogen
    * Patients with stable or declining PSA who have had previous antiandrogen exposure, but are not taking an antiandrogen at the time of registration, must wait at least 6 weeks from the last antiandrogen dose before registration and still demonstrate a stable or falling PSA which is > 4 ng/mL by month 12, in order to be eligible
    * If the PSA is rising and they are on an antiandrogen, formal antiandrogen washout must be performed (4 weeks for flutamide and 6 weeks for bicalutamide and nilutamide with no evidence of a falling PSA after washout)
  * No patients with radiographic progression when compared to available imaging studies performed prior to starting the GNRH agonist/antagonist therapy
* Patients who have measurable disease must have radiographic assessment (at least an abdominal/pelvic CT scan) within 28 days prior to registration
* Non-measurable disease must be assessed (i.e., bone scan) within 42 days prior to registration
* No patients with a history of brain metastases or who currently have treated or untreated brain metastases

  * Patients with clinical evidence of brain metastases must have a brain CT scan or MRI negative for metastatic disease within 56 days prior to registration

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 10 g/dL
* Serum creatinine ≤ 1.5 times the upper limit of normal (ULN) OR creatinine clearance ≥ 60 mL/min
* Bilirubin ≤ 1.5 times ULN (unless documented Gilbert disease)
* AST and ALT < 1.5 times ULN
* Potassium ≥ 3.5 mmol/L
* Patient must have a testosterone value of < 50 ng/dL obtained within 28 days prior to registration
* Patients must have controlled blood pressure defined as systolic blood pressure < 160 mm Hg and diastolic blood pressure < 95 mm Hg

  * Patients with a history of hypertension are eligible provided blood pressure is controlled by anti-hypertensive treatment
* Patients who have partners of child-bearing potential must be willing to use a method of birth control with adequate barrier protection during the study and for 1 week after the last study drug administration
* Must be able to take oral medication without crushing, dissolving, or chewing tablets
* Patients must not have a history of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of abiraterone acetate
* No other prior malignancy is allowed except for any of the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * Adequately treated stage I or II cancer from which the patient is currently in complete remission
  * Any other cancer from which the patient has been disease-free for 5 years
* No patients with active or symptomatic viral hepatitis or chronic liver disease

  * No moderate (Child-Pugh B) or severe (Child-Pugh C) hepatic impairment
* No history of NYHA class III or IV heart failure

  * Patients must have LVEF ≥ 50%
* No known allergies, hypersensitivity, or intolerance to abiraterone acetate, prednisone, or their excipients

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Patients with a history of prior neoadjuvant or adjuvant GNRH agonist/antagonist therapy (related to previous surgery or radiation) are eligible provided they finished this therapy at least two years prior to registration

  * Prior enrollment to SWOG-S0925 (either arm) is not exclusionary
* At least 6 weeks since prior and no concurrent finasteride or dutasteride
* At least 28 days since prior radiotherapy or surgery and recovered
* At least 4 weeks since prior investigational products
* At least 4 weeks since prior flutamide (6 weeks for bicalutamide and nilutamide) with no evidence of a falling PSA

  * No other concurrent oral antiandrogen
* No prior or concurrent cytotoxic chemotherapy or radiopharmaceuticals for prostate cancer
* No prior or concurrent ketoconazole for the treatment of prostate cancer
* Not requiring more than 10 mg a day of prednisone for another medical indication
* Not planning to receive any concurrent cytotoxic chemotherapy, immunotherapy, surgery, or radiotherapy during protocol treatment
* No concurrent hormonal-acting agents, including diethylstilbestrol/DES, aldosterone, PC-SPES, or spironolactone
* No concurrent antifungal medication (e.g., fluconazole or itraconazole)
* No medications that alter cardiac conduction
* No prior Provenge (sipuleucel-T)

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-08-09; Primary Completion 2016-11-29 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W. Flaig, MD, Principal Investigator — University of Colorado, Denver
Locations (205):
- United States (205):
  - NEA Medical Clinic - East Matthews, Jonesboro, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Springdale, Rogers, Arkansas
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Fresno Medical Center, Fresno, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - University of California Davis Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center - Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Oncare Hawaii, Incorporated - Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute, Nampa, Idaho
  - Mountain States Tumor Institute at St. Luke's, Twin Falls, Idaho
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Mid-Illinois Hematology-Oncology Associates at Community Cancer Center, Normal, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - St. Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Hospital Corporation, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas City Cancer Centers - West, Kansas City, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Kansas City Cancer Center - Shawnee Mission, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Hematology-Oncology Clinic, Baton Rouge, Louisiana
  - Cancer Center of Acadiana at Lafayette General Medical Center, Lafayette, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Caritas Holy Family Hospital, Methuen, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute, Flint, Michigan
  - Singh and Arora Hematology Oncology, PC, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Great Lakes Cancer Institute - Lapeer Campus, Lapeer, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Clemens Regional Medical Center, Mount Clemens, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Centers - East, Lee's Summit, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Falck Cancer Center at Arnot Ogden Medical Center, Elmira, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Winthrop University Hospital, Mineola, New York
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Baylor University Medical Center - Houston, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - St. Luke's Texas Cancer Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Rocky Mountain Oncology, Casper, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
http://swog.org/Visitors/Download/Policies/Policy43.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Acetate + Prednisone: Abiraterone, 1,000 mg, oral (on an empty stomach at least 2 hours after or 1 hour before eating); to be taken daily
  Prednisone, 5 mg, oral, 5 mg twice daily
  abiraterone acetate: 1,000 mg, oral (on an empty stomach at least 2 hours after or 1 hour before eating); taken daily
  Prednisone: 5 mg, oral, 5 mg twice daily
Period: Overall Study
Arm/Group | Abiraterone Acetate + Prednisone
Started | 41
Received Protocol Treatment | 40
Completed | 4
Not Completed | 37
Not completed — Lack of Efficacy | 20
Not completed — Other | 9
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: One patient is excluded due to patient not receiving any protocol treatment.
Arm/Group | Abiraterone Acetate + Prednisone
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 66 [39 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 4
  Ethnicity: Not Hispanic/unknown | 36
Testosterone [Median (Full Range); unit: ng/dL] | 12.8 [3.0 to 50.0]
PSA at entry [Median (Inter-Quartile Range); unit: ng/mL] | 23.6 [11.7 to 64.4]
Performance Status [Count of Participants; unit: Participants] — Zubrod Performance Status Scale:
  0= Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. Capable of limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  Participants
    0-1 | 39
    2 | 1
Gleason Score [Count of Participants; unit: Participants] — Pathologists grade prostate cancers using numbers from 1 to 5 based on how much the cells in the cancerous tissue look like normal tissue. This is called the Gleason system.
  If the cancerous tissue looks like normal tissue, a grade of 1 is assigned. If the cancer cells look very abnormal, a grade of 5 is assigned. Grades 2-4 have features in between these extremes.
  Since prostate cancers often have areas with different grades, a grade is assigned to the 2 areas that make up most of the cancer. These 2 grades are added to yield the Gleason score. The highest a Gleason score can be is 10.
  Participants
    2-6 | 3
    7 | 7
    8-10 | 30
Metastasis [Count of Participants; unit: Participants]
  Bone | 37
  Lymph node | 8
  Visceral | 6
Prostate RT [Count of Participants; unit: Participants]
  Yes | 5
  No | 35
Prostatectomy [Count of Participants; unit: Participants]
  Yes | 5
  No | 35
Antiandrogen use [Count of Participants; unit: Participants]
  Yes | 35
  No | 5
PSA status at registration [Count of Participants; unit: Participants]
  Rising level | 34
  Stable/falling level | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Undetectable PSA
Description: undetectable PSA defined as <= 0.2 ng/mL. Patients not responding in the first year were deemed non-responders.
Time Frame: 12 months
Population: All patients who received at least 1 dose of protocol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate + Prednisone
Number analyzed (Participants) | 40
Participants | 5

2. Secondary Outcome: Number of Patients With PSA Partial Response
Description: PSA reduction to < 4 ng/ml, but >0.2 ng/ml
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate + Prednisone
Number analyzed (Participants) | 40
Participants | 13

3. Secondary Outcome: Objective Progression-free Survival
Description: Progression defined as unequivocal progression of disease, progressive disease as defined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), progressive disease as defined by the Prostate Cancer Clinical Trials Working Group bone scan progression criteria, or death due to disease.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abiraterone Acetate + Prednisone
Number analyzed (Participants) | 40
months | 17.5 [8.6 to 25.0]

4. Secondary Outcome: Overall Survival
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abiraterone Acetate + Prednisone
Number analyzed (Participants) | 40
months | 25.8 [15.7 to 25.8]

5. Secondary Outcome: Number of Patients With Toxicity of Abiraterone Acetate
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 3 years
Population: All participants receiving at least some protocol treatment
Measure: Number; unit: Participants
Groups:
- Abiraterone Acetate + Prednisone: Abiraterone: 1,000 mg, oral (on an empty stomach at least 2 hours after or 1 hour before eating); to be taken daily Prednisone: 5 mg, oral, 5 mg twice daily
Arm/Group | Abiraterone Acetate + Prednisone
Number analyzed (Participants) | 40
Participants
  Alanine aminotransferase increased | 2
  Anorexia | 1
  Aspartate aminotransferase increased | 2
  Hyperglycemia | 2
  Hypertension | 2
  Hypokalemia | 2
  INR increased | 1
  Leukocytosis | 1
  Lung infection | 1
  Nausea | 2
  Rectal hemorrhage | 1
  Thromboembolic event | 1
  Vomiting | 2
  Weight gain | 1

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Participants were monitored for toxicity every 2 weeks for the first 3 months, then monthly thereafter or at more frequent intervals appropriate for that participant, as judged by the treating physician.
Arm/Group | Abiraterone Acetate + Prednisone
Serious Adverse Events (participants affected / at risk) | 16/40
Other Adverse Events (participants affected / at risk) | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate + Prednisone (N=40)
Anemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Aortic valve disease (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Retinal detachment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Rectal hemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Lung infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paresthesia (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate + Prednisone (N=40)
Anemia (Blood and lymphatic system disorders) | 12
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 3
Ear and labyrinth disorders-Other (Ear and labyrinth disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Chills (General disorders) | 2
Edema limbs (General disorders) | 8
Fatigue (General disorders) | 15
Pain (General disorders) | 6
Bronchial infection (Infections and infestations) | 2
Infections and infestations-Other (Infections and infestations) | 3
Upper respiratory infection (Infections and infestations) | 4
Bruising (Injury, poisoning and procedural complications) | 4
Fracture (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 10
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 4
Weight gain (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 14
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 4
Nervous system disorders-Other (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 6
Urinary frequency (Renal and urinary disorders) | 3
Pelvic pain (Reproductive system and breast disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3
Surgical and medical procedures-Other (Surgical and medical procedures) | 2
Hot flashes (Vascular disorders) | 11
Hypertension (Vascular disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT01309672/Prot_SAP_002.pdf
  • Informed Consent Form (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT01309672/ICF_001.pdf